CLINICAL TRIAL: NCT02866279
Title: Immediate Postpartum Contraceptive Implant Placement and Breastfeeding Success in Women at Risk for Low Milk Supply: A Non-inferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-6852
Record Dates: First submitted 2016-08-07; First posted 2016-08-15 (Estimated); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Contraception; Breastfeeding; Postpartum Contraception
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Postplacental (Experimental): contraceptive implant placed within 30 minutes of placental delivery
  Interventions: Device: Etonogestrel Contraceptive Implant
- Immediate Postpartum (Experimental): Contraceptive Implant placed 1-3 days postpartum
  Interventions: Device: Etonogestrel Contraceptive Implant
- Delayed (Active Comparator): Contraceptive Implant placed 6 or more weeks postpartum
  Interventions: Device: Etonogestrel Contraceptive Implant

INTERVENTIONS:
Device: Etonogestrel Contraceptive Implant — Women will be randomized to the TIMING of implant placement
  Other Names: Nexplanon

SUMMARY:
The investigators goal is to measure the impact of timing of postpartum contraceptive implant insertion on breastfeeding success and duration and to explore women's experiences with and attitudes towards contraceptive and breastfeeding counseling in the peripartum time period

DETAILED DESCRIPTION:
Immediate postpartum initiation of the etonogestrel contraceptive implant has been proven to decrease rates of rapid, repeat pregnancies. Evidence supports that in healthy women with term infants initiation of the contraceptive implant 1-3 days postpartum does not appear to have any adverse effects on lactogenesis or breastfeeding continuation. However, no high quality study to date has examined the effects of progestin-only contraception in women known to be at risk for low milk supply, including women with a premature delivery, obesity, polycystic ovarian syndrome, diabetes, or a prior history of low milk supply.

The investigators goal is to measure the impact of timing of postpartum contraceptive implant insertion on breastfeeding success and duration. This will be a three-armed randomized non-inferiority study of women who plan to breastfeed, have known risk factors for low milk supply, and who intend to use the contraceptive implant postpartum. Women will be randomized to one of three groups for the timing of contraceptive implant placement: within 30 minutes of placental delivery, 24-72 hours postpartum, or 6 or more weeks postpartum. Women will be assessed at 6 weeks, 3 months and 6 months postpartum. Outcomes will include time to Lactogenesis Stage II, duration and exclusivity of breastfeeding, continuation of and satisfaction with the contraceptive implant, and side effects, including bleeding patterns, associated with the implant.

Findings from this trial will be used by clinicians, hospital systems, and policy makers working to expand access to immediate postpartum implants while supporting women in meeting their breastfeeding goals.

ELIGIBILITY:
Inclusion Criteria:

* Live pregnancy of at least 24 weeks gestation
* Intention to use a contraceptive implant postpartum
* 17 years of age or older
* English or Spanish speaking
* Admission to Labor and Delivery with a plan for delivery (women in both latent and active labor will be eligible)
* The presence of at least one of the following conditions known to be a risk factor for low milk supply:

  * Expected delivery prior to 34 weeks
  * Obesity (pre-pregnancy BMI >35)
  * Polycystic Ovarian Syndrome
  * Diabetes (gestational or pre-gestational)
  * Self-reported difficulty with low milk supply in past

Exclusion Criteria:

* Not English or Spanish speaking
* Allergy or Contraindication to contraceptive implant

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 155 (Actual)
Dates: Start 2016-11; Primary Completion 2021-04-07 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Levi, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Gurtcheff SE, Turok DK, Stoddard G, Murphy PA, Gibson M, Jones KP. Lactogenesis after early postpartum use of the contraceptive implant: a randomized controlled trial. Obstet Gynecol. 2011 May;117(5):1114-1121. doi: 10.1097/AOG.0b013e3182165ee8. PMID 21508750
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Postplacental | Immediate Postpartum | Delayed
Started | 51 | 52 | 52
Completed | 51 | 52 | 52
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Postplacental | Immediate Postpartum | Delayed | Total
Number analyzed (Participants) | 51 | 52 | 52 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (4.5) | 27 (4.6) | 27 (4.8) | 27 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 52 | 52 | 155
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 32 | 31 | 95
  Not Hispanic or Latino | 14 | 17 | 18 | 49
  Unknown or Not Reported | 5 | 3 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 18 | 22 | 65
  White | 9 | 8 | 6 | 23
  More than one race | 17 | 24 | 24 | 65
  Unknown or Not Reported | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Breastfeeding at 6 Months
Description: Exclusive Breastfeeding at 6 months
Time Frame: 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Postplacental | Immediate Postpartum | Delayed
Number analyzed (Participants) | 51 | 52 | 52
Participants | 6 | 4 | 6

2. Primary Outcome: Time to Lactogenesis Stage II
Description: Difference in time to Lactogenesis Stage II
Time Frame: 1-5 days postpartum
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Postplacental | Immediate Postpartum | Delayed
Number analyzed (Participants) | 51 | 52 | 52
hours | 66.9 (27.2) | 62.1 (29.0) | 57.3 (21.7)

3. Secondary Outcome: Vaginal Bleeding
Description: Number of Participants that reported heavy bleeding at 6 months postpartum
Time Frame: 0-6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Postplacental | Immediate Postpartum | Delayed
Number analyzed (Participants) | 51 | 52 | 52
Participants | 7 | 6 | 4

4. Secondary Outcome: Satisfaction With Contraceptive Implant
Description: Satisfaction on a 1-10 scale (10 being highly satisfied) at 6 months postpartum
Time Frame: 0-6 months postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Postplacental | Immediate Postpartum | Delayed
Number analyzed (Participants) | 51 | 52 | 52
score on a scale | 8.41 (2.01) | 8.14 (2.47) | 8.69 (1.60)

ADVERSE EVENTS:
Time Frame: Every 3 months from initiation to 6 months post-partum
Arm/Group | Postplacental | Immediate Postpartum | Delayed
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/51 | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02866279/Prot_SAP_000.pdf